CLINICAL TRIAL: NCT00527020
Title: Single-Blind, Randomised, Placebo-controlled First Time in Human Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Oral Escalating Doses of GSK1018921 in Healty Volunteers and a Randomized, Double-blind, Double Dummy, Placebo Controlled, Three-way Crossover Study in a Separate Cohort of Healthy Volunteers to Test the Effect of Single Doses of GSK1018921 and Nicotine on qEEG and MMN in Healthy Volunteers
Brief Title: First Time in Human Study With GSK1018921
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: GT1109727
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia
Keywords: qEEG,; GlyT-1 inhibitor,; ERP; GSK1018921,; FTIH,; schizophrenia,; single-dose,; healthy volunteers,; MMN,
MeSH Terms: conditions — Schizophrenia | interventions — GSK 1018921; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part A: Subjects receiving treatment in cohort A (Experimental): Eligible subjects will be randomized to receive GSK101892 and placebo. Subjects will receive escalated doses of GSK101892 with a starting dose of 0.5 milligrams. Each subject will receive no more than 4 doses of GSK1018921 in a maximum of 5 dosing sessions. Within each cohort, each session will be separated by a washout period of at least 7 days.
  Interventions: Drug: GSK1018921; Drug: Nicotine Lozenges; Drug: Placebo
- Part A: Subjects receiving treatment in cohort B (Experimental): Eligible subjects will be randomized to receive GSK101892 and placebo. Subjects will receive escalated doses of GSK101892 with a starting dose of 0.5 milligrams. Each subject will receive no more than 4 doses of GSK1018921 in a maximum of 5 dosing sessions. Within each cohort, each session will be separated by a washout period of at least 7 days.
  Interventions: Drug: GSK1018921; Drug: Nicotine Lozenges; Drug: Placebo
- Part A: Subjects receiving treatment in cohort C (Experimental): Eligible subjects will be randomized to receive GSK101892 and placebo. Subjects will receive escalated doses of GSK101892 with a starting dose of 0.5 milligrams. Each subject will receive no more than 4 doses of GSK1018921 in a maximum of 5 dosing sessions. Within each cohort, each session will be separated by a washout period of at least 7 days.
  Interventions: Drug: GSK1018921; Drug: Nicotine Lozenges; Drug: Placebo
- Part B: Subjects in 5 period crossover period (Experimental): Eligible subjects (first 14 subjects) will be randomized to one of the following 14 sequences as a 5 period crossover with sequences; LMNOQ, MNOLQ, NOLMQ, OLMNQ, ONMLQ, NMLOQ, MLONQ, LONMQ, LNMOQ, NMOLQM MOLNQ, OLNMQ, OMNLQ and MNLOQ) (L= 80 milligrams GSK1018921 given in fasted state, M= 200 milligrams GSK1018921 given in fasted state, N= nicotine lozenge, O= placebo and Q= 80 milligrams GSK1018921 in fed state).
  Interventions: Drug: GSK1018921; Drug: Nicotine Lozenges; Drug: Placebo
- Part B: Subjects in 4 period crossover period (Experimental): Eligible subjects (last 7 subjects) will be randomized to one of the following 7 sequences as a 4 period crossover with sequences; NLOM, LOMN, OLNM, LNMO, NMOL, MOLN, and MNLO.
  Interventions: Drug: GSK1018921; Drug: Nicotine Lozenges; Drug: Placebo

INTERVENTIONS:
Drug: GSK1018921 — GSK1018921 will be supplied as 0.5, 5, 10 and 40 milligrams coated tablets.
Drug: Nicotine Lozenges — Nicotine Lozenges will be supplied as 4 milligrams lozenges.
Drug: Placebo — Placebo tablets will be given to the subjects.

SUMMARY:
GSK1018921 is a new drug under development for the treatment of schizophrenia. GSK1018921 differs from other available drugs in its mode of action and it is assumed that it may have an effect in the treatment of so-called positive symptoms such as hallucinations and negative symptoms such as lack of drive. No clinical studies have been conducted with GSK1018921 in humans until now. This is the first study where this compound is administered to humans; the study has 2 parts: Part A is a dose escalation study, Part B is a pharmacodynamic portion in a separate group of healthy smoker volunteers.

DETAILED DESCRIPTION:
Single-Blind, Randomised, Placebo-Controlled First Time in Human Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Oral Escalating Doses of GSK1018921 in Healthy Volunteers and to assess the effect of a single dose of GSK1018921 on quantitative EEG and Mismatch Negativity in a separate cohort of healthy smoker volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers as determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, cardiac monitoring.
* For Part B, smokers.

Exclusion Criteria:

* Part A: Smokers, any subject who takes any prescribed or non-prescribed medication/vitamins specified as prohibited in the protocol, substance abuse, clinically significant disease as determined by a responsible physician.
* Part B: Non-Smokers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2007-08-10 (Actual); Primary Completion 2008-07-12 (Actual); Study Completion 2008-07-12 (Actual)

PRIMARY OUTCOMES:
Part A:Safety pre-dose-8-15days post dose Tolerability,PK of single escalating doses. Part B: PD effects of single doses of GSK1018921 and nicotine on Quantitative Electroencephalography and MisMatch Negativity in smokers. | pre-dose-8-15days post dose

SECONDARY OUTCOMES:
Part A:Characterise single-dose PD with Bond-Lader Visual analogue Scale,Profile of Mood State,Glycine levels.Part B:Safety pre-dose-8-15 days post dose,Tolerability,PK of single escalating doses.Amplitude and latency of P300, Effects on P50 suppression | pre-dose-8-15 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- [Background] Ouellet D, Sutherland S, Wang T, Griffini P, Murthy V. First-time-in-human study with GSK1018921, a selective GlyT1 inhibitor: relationship between exposure and dizziness. Clin Pharmacol Ther. 2011 Oct;90(4):597-604. doi: 10.1038/clpt.2011.154. Epub 2011 Aug 24. PMID 21866096
- See also: Results for study GT1109727 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/GT1109727?search=study&study_ids=GT1109727#rs